CLINICAL TRIAL: NCT05058560
Title: Tislelizumab in Addition to Bronchial Arterial Chemoembolization in Patients with Non-Small-Cell Lung Cancer -- a Single-arm Phase II Trial
Brief Title: Tislelizumab in Addition to BACE in Patients with NSCLC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The First Affiliated Hospital of Zhengzhou University (Other)
Responsible Party: Principal Investigator, Xuhua Duan, Associate Professor, The First Affiliated Hospital of Zhengzhou University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20210831
Record Dates: First submitted 2021-08-31; First posted 2021-09-27 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: NSCLC
Keywords: BACE; PD-1
MeSH Terms: interventions — tislelizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- BACE+Tislelizumab (Experimental): BACE was performed on the first day of the first cycle, and the first 200 mg of tislelizumab was given 3-5 days later.
  Interventions: Drug: Tislelizumab

INTERVENTIONS:
Drug: Tislelizumab — tislelizumab, 200 mg IV Q3W, up to one year.
  Other Names: Bronchial artery chemoembolization (BACE)

SUMMARY:
This is a single-arm phase II trial to determine the efficacy and safety of Tislelizumab in addition to bronchial arterial chemoembolization in stage III-Ⅳ NSCLC patients who failed, refused or ineligible to receive standard treatments.

DETAILED DESCRIPTION:
Bronchial artery chemoembolization (BACE) is a technique of drug delivery and embolization performed via injecting anti-tumor drugs with drug carriers and implanting the embolization agents into the tumor feeding artery, promoting the clinical outcomes of patients and providing a palliative treatment option for patients with NSCLC. while the short-term effect of BACE is good, it is easy to relapse and metastasize.

The rapid development of immunotherapy checkpoint inhibitors represented by PD-1/L1 monoclonal antibody has changed the treatment pattern of NSCLC. The publication of early research data repeatedly verified the long-term survival benefit characteristics of PD-1/L1 in NSCLC.

Tislelizumab is an investigational humanized IgG4 monoclonal antibody with high affinity and binding specificity for PD-1. Tislelizumab was engineered to minimize binding to FcγR on macrophages in order to limit antibody-dependent phagocytosis, a potential mechanism of resistance to anti-PD-1 therapy. Tislelizumab in combination with platinum-based chemotherapy as first-line treatment for advanced SCLC and NSCLC, including nsq-NSCLC, resulted in robust responses in a phase 2 study (BGB-A317-206 [NCT03432598]), In phase 3 study, addition of tislelizumab to chemotherapy resulted in significantly improved progression-free survival (PFS) compared with chemotherapy alone in patients with stage IIIB or IV squamous NSCLC (RATIONALE 307; BGB-A317-307 [NCT03594747]) and nsq-NSCLC (RATIONALE 304; BGB-A317-304 [NCT03663205]). Second-and third-line tislelizumab monotherapy prolonged OS in the ITT and PD-L1 ≥ 25% populations vs docetaxel in patients with advanced NSCLC(RATIONALE 303; BGB-A317-303 [NCT03358875]). China NMPA have approved for tislelizumab + chemotherapy for 1L NSCLC.

This trial is designed to determine the efficacy and safety of Tislelizumab in addition to Bronchial Arterial Chemoembolization in stage III-Ⅳ NSCLC patients who failed, refused or ineligible to receive standard treatments.

ELIGIBILITY:
Inclusion Criteria:

1. Patient age between 18 and 75
2. Signed Informed Consent Form.
3. Confirmed TNM stage is III-Ⅳ of NSCLC ，and failed, refused or assessed ineligible to receive conventional treatments (surgery, chemoradiotherapy, Chemotherapy)；
4. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 1
5. Adequate hematologic and end-organ function.
6. Expected life span > 3 months.
7. Be able to provide fresh or archival tumor tissues for PD-L1 expression in tumor cells

Exclusion Criteria:

1. Prior therapies of docetaxel or treatment targeting PD-1, PD-L1 or CTLA-4.
2. Prior therapies of interventional therapy (I seeds implantation, Ablation, BACE).
3. Harboring EGFR sensitizing mutation or ALK gene translocation
4. History of interstitial lung disease, non-infectious pneumonitis or participants with significantly impaired pulmonary function, or who require supplemental oxygen at baseline.
5. With uncontrollable pleural effusion, pericardial effusion, or clinically significant ascites requiring interventional treatment.
6. Symptomatic central nervous system metastasis
7. Known HIV infection, participants with untreated chronic hepatitis B, active vaccination treatment.
8. Prior allogeneic stem cell transplantation or organ transplantation
9. Active autoimmune diseases or history of autoimmune diseases that may relapse.
10. With conditions requiring systemic treatment with either corticosteroids (>10 mg daily prednisone or equivalent) or other immunosuppressive medications
11. Known to be hypersensitive to contrast agent;
12. Pregnant or breastfeeding women;
13. Other protocol defined Inclusion/Exclusion criteria may apply

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2025-02-04 (Actual); Study Completion 2025-02-15 (Actual)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | Time from the first BACE treatment to either radiological progression or death or up to 12 months
  Time from the first BACE treatment to either radiological progression or death

SECONDARY OUTCOMES:
Objective response rate (ORR) | 2, 4, 6 months after the first BACE treatment, up to death or 12 months
  Proportion of patients with reduction in stable in tumor burden of a predefined amount
Disease control rate (DCR) | 2, 4, 6 months after the first BACE treatment, up to death or 12 months
  Proportion of patients with reduction or keeping in stable in tumor burden of a predefined amount
Overall survival (OS) | 1 years or more
  Time from the first BACE treatment to death from any cause or the end of the study
Quality of life score (EORTC, QLQ-30) | Every two months after treatment when the patient was assessed complete response; every month after treatment when assessed partial response, stable disease or progressive disease; up to progressive disease after the second treatment or within 12 months
  Changes of quality of life score; using the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-30) Scores

CONTACTS AND LOCATIONS:
Overall Officials: Xuhua Duan, Principal Investigator — Zhengzhou University - First Affiliated Hospital
Locations (1):
- The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Hennan, China